CLINICAL TRIAL: NCT00005914
Title: Genetics of Recurrent Early-Onset Depression
Acronym: GenRED
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Douglas F. Levinson, Principle Investigator, Stanford University
Other Study IDs: R01MH061686-01 (NIH); R01MH061686-01 (NIH); R01MH060912 (NIH); R01MH059552 (NIH); R01MH059541 (NIH); R01MH059542 (NIH); R01MH061686 (NIH); R01MH060866 (NIH); DNBBS 7G-GRR
Record Dates: First submitted 2000-06-15; First posted 2000-06-16 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Depression
Keywords: Depression; Depressive Disorder; Family; Genes; Genetic Techniques; Genetics; Linkage (Genetics); Nuclear Family; Recurrence; Severity of Illness Index
MeSH Terms: conditions — Depression; Depressive Disorder; Recurrence

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood specimens were submitted to the NIMH repository at the Rutgers University Cell and DNA Repository.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Probands and family members: Individuals with major depressive disorder who meet study criteria, and members of their families. No intervention. This is a genetic study only.

SUMMARY:
This nationwide study will create a DNA collection to permit qualified scientists to search for depression-related genes.

More than 750 families with at least two siblings who have experienced major depression are needed for the study. Participants will be interviewed about psychiatric and family history, and will be asked to provide a small blood specimen. The identification of predisposing genes can lead to greater understanding of the brain mechanisms involved in severe depression which can in turn lead to the discovery of new treatments.

A Certificate of Confidentiality from the federal government ensures that all information will be strictly confidential. Blood specimens are identified only by code number (not by name).

Reimbursement is provided.

DETAILED DESCRIPTION:
Studies of patterns of major depression in families suggest that 50 to 70% of the predisposition to major depression is caused by genes. People with recurrent depression and earlier ages of onset have more relatives with depression. There are probably at least several interacting genes, rather than a single gene as in some disorders. The identification of predisposing genes is likely to lead to greater understanding of the brain mechanisms involved in severe depression. This could lead to the discovery of new treatments.

This study will create a DNA collection to permit qualified scientists to search for depression-related genes. More than 750 families with at least two siblings who have experienced major depression are needed for the study.

Participants in this study will be interviewed about psychiatric and family history, and will be asked for a small blood specimen. Interviews can be conducted in person or by telephone. For telephone interviews, blood sample collection will be arranged at a location and time convenient for the participant. Participants will also be asked for help in inviting other family members to participate. No family member will be contacted without the permission and assistance of another participating family member.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00260182

ELIGIBILITY:
Inclusion Criteria:

* Families that have at least TWO ADULT SIBLINGS (brother/brother; sister/sister; brother/sister) who have experienced major depression.
* Depression must be RECURRENT (more than one episode).
* Depression must have started at age 30 or less in one sibling, and at age 40 or less in the other sibling.

Exclusion Criteria:

* Participants cannot have Bipolar I (manic-depressive) disorder or schizophrenia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Probands will have major depressive disorder meeting the eligibility criteria described below.
Sampling Method: Non-Probability Sample
Enrollment: 2533 (Actual)
Dates: Start 1999-10; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Major depressive disorder | One patient interview session (typically 2 hours), and blood draw (10-20 minutes)
  Participants will attend an interview regarding personal and family history of psychiatric disorders, and give a blood specimen. Genotypes from blood samples will be studied for genetic linkage (within families) with the presence of major depressive disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Myrna Weissman, Principal Investigator — Columbia University; J R DePaulo, Principal Investigator — Johns Hopkins University; William Scheftner, Principal Investigator — Rush University Hospital; Raymond Crowe, Principal Investigator — University of Iowa; Douglas Levinson, Principal Investigator — University of Pennsylvania; George Zubenko, Principal Investigator — University of Pittsburgh
Locations (6):
- United States (6):
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Univ of Iowa Hosp and Clinic, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - New York State Psychiatric Institute / Columbia Univ, New York, New York
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Univ of Pittsburgh / Western Psychiatric Inst and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Web site for New York Psychiatric Institute — http://nyspi.org
- See also: Web site for University of Iowa — http://www.medicine.uiowa.edu/psychiatry/